CLINICAL TRIAL: NCT00340587
Title: Human Sperm Binding to Transgenic Mouse Eggs
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997039; OH97-DK-N039
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-02-24

CONDITIONS: Fertilization
Keywords: Zona Pellucida; Human Eggs; ZP1, ZP2, ZP3; Fertilization

SUMMARY:
At fertilization, the binding of sperm to the zona pellucida induces the acrosome reaction releasing lytic enzymes that facilitate the passage of the sperm through the zona. The sperm then fuses with the egg's plasm membrane and enters the egg's cytoplasm. The zona pellucida, an extracellular matrix composed of three glycoproteins (ZP1, ZP2, ZP3), mediates the species-specific binding of sperm to egg. Although homologous proteins are present in mouse and humans, human sperm will not bind to the mouse zona pellucida and when the zona pellucida is experimentally removed, human sperm will not bind or fuse to the mouse egg's plasm membrane. We have created transgenic mouse lines that express one or more human zona proteins. We wish to determine if human sperm will bind to these chimeric zonae and if this binding will induce the human sperm acrosome reaction. Sperm and devitalized eggs will be collected by collaborating institution(s) under protocols and consent forms approved by that institution's IRB. Only procedures already being performed on subjects for diagnostic or treatment purposes will be used.

DETAILED DESCRIPTION:
At fertilization, the binding of sperm to the zona pellucida induces the acrosome reaction releasing lytic enzymes that facilitate the passage of the sperm through the zona. The sperm then fuses with the egg s plasma membrane and enters the egg s cytoplasm. The zona pellucida, an extracellular matrix composed of three or four glycoproteins, mediates the species-specific binding of sperm to egg. Although homologous proteins are present in mouse and humans, human sperm will not bind to the mouse zona pellucida and when the zona pellucida is experimentally removed, human sperm will not bind or fuse to the mouse egg's plasma membrane. We have established transgenic mouse lines that express one or more human or rat zona proteins. We wish to determine if human sperm will bind to these chimeric zonae and if this binding will induce the human sperm acrosome reaction. Sperm and devitalized eggs will be collected by collaborating institution(s) under protocols and consent forms approved by that institution's IRB. Alternatively, anonymous fertile human sperm will be obtained from a commercial sperm bank using a donor consent agreement. Only procedures already being performed on subjects for diagnostic or treatment purposes will be used.

ELIGIBILITY:
* INCLUSION CRITERIA:

Without regard to ethnic/race background, all subjects will be men and women over the age of 18 who are neither mentally retarded nor disabled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1997-05-02; Study Completion 2016-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Jurrien Dean, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rankin T, Dean J. The molecular genetics of the zona pellucida: mouse mutations and infertility. Mol Hum Reprod. 1996 Nov;2(11):889-94. doi: 10.1093/molehr/2.11.889. PMID 9237231
- [Background] Rankin T, Familari M, Lee E, Ginsberg A, Dwyer N, Blanchette-Mackie J, Drago J, Westphal H, Dean J. Mice homozygous for an insertional mutation in the Zp3 gene lack a zona pellucida and are infertile. Development. 1996 Sep;122(9):2903-10. doi: 10.1242/dev.122.9.2903. PMID 8787763
- [Background] Epifano O, Liang LF, Familari M, Moos MC Jr, Dean J. Coordinate expression of the three zona pellucida genes during mouse oogenesis. Development. 1995 Jul;121(7):1947-56. doi: 10.1242/dev.121.7.1947. PMID 7635043